CLINICAL TRIAL: NCT03709771
Title: Novel Mechanisms and Predictors of VEGF Receptor Inhibitor- or Immune Checkpoint Inhibitor-Associated Hypertension and Cardiovascular Disease
Status: Terminated | Type: Observational
Why Stopped: Study terminated due to unmet targeted accrual goals with only 2 subjects accrued out of 80 planned due to COVID-19 and the PI on the grant leaving VUMC in October 2021.
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Joshua Beckman, Professor, Vanderbilt University Medical Center
Other Study IDs: 181796
Record Dates: First submitted 2018-10-15; First posted 2018-10-17 (Actual); Results first posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2023-04

CONDITIONS: Renal Cell Carcinoma; Hypertension; Melanoma; Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Hypertension; Melanoma; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- VEGF inhibitor alone
  Interventions: Diagnostic Test: Ambulatory Blood Pressure Measurement
- Immune Checkpoint Inhibitor (ICI) alone
  Interventions: Diagnostic Test: Ambulatory Blood Pressure Measurement
- Combination (VEGF inhibitor + ICI, or combination of ICI)
  Interventions: Diagnostic Test: Ambulatory Blood Pressure Measurement
- No treatment
  Interventions: Diagnostic Test: Ambulatory Blood Pressure Measurement

INTERVENTIONS:
Diagnostic Test: Ambulatory Blood Pressure Measurement — Baseline: Subjects will undergo an abbreviated physical exam, review changes in medical history since last oncology visit, blood collection, urine collection, blood pressure and heart rate in triplicate, baseline and hyperemic digital velocity time interval (VTI) using pulse amplitude tonometry, cubital vein endothelial cell harvest, and ambulatory 24 blood pressure measurement.
  Follow-up Visit (approx 1 month after starting treatment): Review changes in medications and any medical events that happened since the last visit, an abbreviated physical exam, blood collection, urine collection, blood pressure and heart rate in triplicate, baseline and hyperemic velocity time interval (VTI), digital pulse amplitude tonometry, endothelial cell harvest, and ambulatory 24 blood pressure.

SUMMARY:
The purpose of this study is to understand the effect of vascular endothelial growth factor tyrosine kinase (VEGF) inhibitor, immune checkpoint-inhibitor (ICI), and combination treatment on blood pressure and blood vessel function.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 40 - 75 years old
* Diagnosis of cancer
* Receiving VEGF inhibitor, ICI, or combination (VEGF inhibitor + ICI or combination ICI) treatment, or not receiving any treatment.
* Normal blood pressure or blood pressure treated to < 140/90 mm Hg with ≤2 antihypertensive medications

Exclusion Criteria:

* Presence of peripheral artery disease
* History of a heart attack within 1 year
* History of a stroke within 1 year
* Diabetes
* Life expectancy < 3 months
* Women who are pregnant
* Women who are nursing

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with cancer that will be receiving VEGF inhibitor, ICI, or combination (VEGF inhibitor plus ICI or combination ICI treatment), or not receiving any treatment.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Beckman, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | VEGF Inhibitor Alone | Immune Checkpoint Inhibitor (ICI) Alone | Combination (VEGF Inhibitor + ICI, or Combination of ICI) | No Treatment
Started | 0 | 1 | 1 | 0
Completed | 0 | 1 | 0 | 0
Not Completed | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Data analysis was not completed because only one participant completed the study and disclosing data could violate privacy interests.
Groups:
- Total: Total of all reporting groups
Arm/Group | VEGF Inhibitor Alone | Immune Checkpoint Inhibitor (ICI) Alone | Combination (VEGF Inhibitor + ICI, or Combination of ICI) | No Treatment | Total
Number analyzed (Participants) | 0 | 1 | 1 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 | 0 |  | 0
  Between 18 and 65 years |  | 0 | 1 |  | 1
  >=65 years |  | 1 | 0 |  | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 1 | 0 |  | 1
  Male |  | 0 | 1 |  | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 0 | 0 |  | 0
  Not Hispanic or Latino |  | 1 | 1 |  | 2
  Unknown or Not Reported |  | 0 | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0 |  | 0
  Asian |  | 0 | 0 |  | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0 |  | 0
  Black or African American |  | 0 | 1 |  | 1
  White |  | 1 | 0 |  | 1
  More than one race |  | 0 | 0 |  | 0
  Unknown or Not Reported |  | 0 | 0 |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Blood Pressure
Description: Mean 24 hour blood pressure from ambulatory 24 hour recording
Time Frame: Baseline and 1 month
Population: as for baseline characteristics
Arm/Group | VEGF Inhibitor Alone | Immune Checkpoint Inhibitor (ICI) Alone | Combination (VEGF Inhibitor + ICI, or Combination of ICI) | No Treatment
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Ratio of Post-treatment to Pre-treatment Change in Digital Pulse Amplitude
Description: Digital pulse amplitude will be measured using peripheral artery tonometry
Time Frame: Baseline and 1 month
Population: as for baseline characteristics
Arm/Group | VEGF Inhibitor Alone | Immune Checkpoint Inhibitor (ICI) Alone | Combination (VEGF Inhibitor + ICI, or Combination of ICI) | No Treatment
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from baseline to 1 month.
Description: There were no participants in the other two arms (VEGF alone and no treatment) and therefore there were no participants at risk in those arms.
Arm/Group | VEGF Inhibitor Alone | Immune Checkpoint Inhibitor (ICI) Alone | Combination (VEGF Inhibitor + ICI, or Combination of ICI) | No Treatment
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1 | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1 | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1 | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-12-13): https://cdn.clinicaltrials.gov/large-docs/71/NCT03709771/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-30): https://cdn.clinicaltrials.gov/large-docs/71/NCT03709771/SAP_001.pdf